CLINICAL TRIAL: NCT03340818
Title: Bone Marrow Concentrate Intradiscal Injection for Chronic Discogenic Low Back Pain: A Double-Blind, Placebo Controlled Trial
Brief Title: Bone Marrow Concentrate Intradiscal Injection for Chronic Discogenic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: APM Spine and Sports Physicians (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMC-1788
Record Dates: First submitted 2017-11-02; First posted 2017-11-14 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2020-01

CONDITIONS: Discogenic Pain
Keywords: Low back pain, bone marrow concentrate, disc degeneration
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind placebo controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and PA providing follow up care and assessing data from ODI, VAS etc will be blinded. Physician performing procedure will not be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone Marrow Concentrate (Experimental): Patients in this group will receive injection of autologous bone marrow concentrate into the suspected painful intervertebral discs.
  Interventions: Other: Bone Marrow Concentrate
- Placebo Group (Sham Comparator): Patients in this group will receive an injection of normal saline dorsal to the transverse process. The bone marrow aspiration will be simulated for these patients.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Bone Marrow Concentrate — Bone marrow concentrate is bone marrow harvested from the iliac crest and minimally processed in a centrifuge. It is then injected into the suspected painful disc (s) using fluoroscopic guidance
  Arms: Bone Marrow Concentrate
Other: Placebo — Injection of normal saline dorsal to the transverse process after sham bone marrow aspiration
  Arms: Placebo Group

SUMMARY:
A double-blind, placebo-controlled study to determine the efficacy of intradiscal injection of bone marrow concentrate on discogenic low back pain.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled study to determine the efficacy of intradiscal injection of bone marrow concentrate on discogenic low back pain. The treatment will be a single injection of autologous bone marrow concentrate into suspected painful disc(s) based upon either prior discography or combination of imaging and exclusion of other anatomic structural sources of pain. The placebo treatment will be an intramuscular injection of normal saline directly dorsal to the transverse process at each suspected level. Outcomes will be measured using VAS and ODI. The primary outcome will be the percentage of patients in the treatment group vs control group at 6 months post-procedure, categorized as a clinical success defined by at least 50% relief of pain. Secondary outcomes will be comparison of success rates at 3 and 12 months, percentage of patients in the two groups with greater than 30% improvement in ODI at 3, 6 and 12 months, Global perceived index at 3, 6, 12 months. Medication log and adjunctive treatments will be recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain for more than 6 months w/ low back component greater than leg pain.
* Average pain of at lest 40/100 on VAS pre-procedure.
* Inadequate response to at least 6 months of conservative care including medication, physical therapy and/or spinal injection
* Advanced imaging of MRI or CT demonstrating abnormal disc pathology
* Presumed lumbar disc pain based on either positive discogram or patient must have MRi findings of either high intensity zone and/or Type 1 or 2 Modic endplate changes, or exclusion of other sources of pain.
* Having provided informed consent

Exclusion Criteria:

* Active moderate to severe lumbar radiculopathy
* Negative discogram
* Very severe decrease in disc height at planned injection level (disc height of less than 1/3 expected)
* Active infection
* Moderate to severe anemia, thrombocytopenia or leukopenia
* Spinal fracture within the past 6 months
* Severe psychological illness
* Inability to consent to the procedure due to cognitive issues
* Prior surgery at a level considered to be the source of pain
* Lumbar surgery within the past 6 months
* Women who are pregnant or breast feeding
* Prior intradiscal therapeutic injection or procedure
* Severe uncontrolled renal, hepatic, hematologic, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurological disease or any medical condition which would make the subject unsuitable for this study.
* Inflammatory arthritis
* Any cancer within the past 5 years, except basal cell or squamous cell skin cancer
* Intradural disc herniation
* Coagulopathy preventing spinal injection
* Inability to stop anticoagulants other than aspirin due to other medical issues
* Exceeds 30 mg morphine equivalent per day of opioid use.
* A history of alcohol or drug abuse within the past 5 years.
* Use of any investigational drug within the past 30 days.
* Steroid injection in the spine within the past 30 days.
* Discography within the last 21 days
* A known allergy or sensitivity to heparin or citrate (used for processing BMC)
* Pending litigation involving the subject's back pain.
* Active worker's compensation claim
* Central stenosis at a level to be injected with an AP diameter less than or equal to 5 mm
* Severe anaphylactic/anaphylactoid reaction to any of the medications used. (If a patient does have a mild or moderate allergy to any of the medications used in the procedure or prior anaphylactic/anaphylactoid reaction to any food or drug, they will be given prednisone 50 mg PO 13, 7, and 1 hour prior to the procedure and diphenhydramine 50mg PO 1 hour prior to the procedure.)
* In order to mitigate any economic risk, a patient without adequate medical insurance coverage for any subsequent tests or procedures deemed clinically necessary will be excluded. BMC is an autologous blood product with multiple clinical uses. Intradiscal administration should not preclude insurance coverage for any subsequent medical issues that might develop pertaining to the intradiscal injection itself or the BMC

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2024-08-07 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Pain relief treatment vs placebo group 50% | 6 months
  Pain reduction of at least 50% at 6 months post-procedure using Visual Analog Scale (VAS) as indicators of pain relief. A reduction in the VAS of at least 50% from baseline is considered successful. VAS of 10 is considered "worst pain imaginable" and VAS of 0 is no pain at all.
Functional improvement vs Placebo group 50% | 6 months
  Functional improvement of at least 50% at 6 months post-procedure using the Oswestry Disability Index (ODI). A reduction of at least 50% in the Oswestry Disability Index is considered successful. The lower the ODI score, the less impact the pain has on a patients daily functioning.

SECONDARY OUTCOMES:
Pain relief treatment vs placebo group 50% | 3 months, 12 months
  Pain reduction of at least 50% will be assessed at 3 and 12 months post-procedure using the Visual Analog Scale (VAS). A reduction of VAS score at 3 and 12 months of at least 50% of baseline will be considered successful. A score of 10 is the "worst pain imaginable" and a score of 0 is no pain at all.
Pain relief treatment vs placebo 30% | 3, 6, 12 months
  Pain reduction of at least 30% at 3, 6, 12 months post-procedure using the Visual Analog Scale (VAS). A decrease in score of at least 30% will be considered successful. A score of 10 is "the worst pain imaginable" and a score of 0 is no pain at all.
Functional improvement treatment vs placebo 50% | 3 months, 12 months
  Improvement in daily functioning of at least 50% from baseline using the Oswestry Disability Index (ODI). A decrease in score of ODI of at least 50% will be considered successful.
Functional improvement treatment vs placebo 30% | 3 months, 12 months
  Improvement in daily functioning of at least 30% from baseline using the Oswestry Disability Index (ODI). A reduction in score by 30% is considered successful

OTHER OUTCOMES:
Medication usage | 12 months
  Medication log of use of pain medications pre-procedure vs post-procedure will be assessed to determine if less medication has been taken since the procedure when compared with pre-procedure.
Adjunct therapy | 12 months
  Log of any adjunctive therapies post procedure

CONTACTS AND LOCATIONS:
Overall Officials: David S Levi, MD, Principal Investigator — Jordan Young Institute; Scott I Horn, DO, Study Chair — Jordan Young Institute; Josh Levin, MD, Study Chair — Stanford University; Sara A Tyszko, PA-C, Study Chair — Jordan Young Institute
Locations (1):
- Jordan Young Institute, Virginia Beach, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schwarzer AC, Aprill CN, Derby R, Fortin J, Kine G, Bogduk N. The prevalence and clinical features of internal disc disruption in patients with chronic low back pain. Spine (Phila Pa 1976). 1995 Sep 1;20(17):1878-83. doi: 10.1097/00007632-199509000-00007. PMID 8560335
- [Background] Fritzell P, Hagg O, Wessberg P, Nordwall A; Swedish Lumbar Spine Study Group. 2001 Volvo Award Winner in Clinical Studies: Lumbar fusion versus nonsurgical treatment for chronic low back pain: a multicenter randomized controlled trial from the Swedish Lumbar Spine Study Group. Spine (Phila Pa 1976). 2001 Dec 1;26(23):2521-32; discussion 2532-4. doi: 10.1097/00007632-200112010-00002. PMID 11725230
- [Background] Hanley EN Jr, David SM. Lumbar arthrodesis for the treatment of back pain. J Bone Joint Surg Am. 1999 May;81(5):716-30. doi: 10.2106/00004623-199905000-00015. No abstract available. PMID 10360702
- [Background] Peng B, Wu W, Hou S, Li P, Zhang C, Yang Y. The pathogenesis of discogenic low back pain. J Bone Joint Surg Br. 2005 Jan;87(1):62-7. PMID 15686239
- [Background] Coppes MH, Marani E, Thomeer RT, Groen GJ. Innervation of "painful" lumbar discs. Spine (Phila Pa 1976). 1997 Oct 15;22(20):2342-9; discussion 2349-50. doi: 10.1097/00007632-199710150-00005. PMID 9355214
- [Background] Freeman BJ, Fraser RD, Cain CM, Hall DJ, Chapple DC. A randomized, double-blind, controlled trial: intradiscal electrothermal therapy versus placebo for the treatment of chronic discogenic low back pain. Spine (Phila Pa 1976). 2005 Nov 1;30(21):2369-77; discussion 2378. doi: 10.1097/01.brs.0000186587.43373.f2. PMID 16261111
- [Background] Barendse GA, van Den Berg SG, Kessels AH, Weber WE, van Kleef M. Randomized controlled trial of percutaneous intradiscal radiofrequency thermocoagulation for chronic discogenic back pain: lack of effect from a 90-second 70 C lesion. Spine (Phila Pa 1976). 2001 Feb 1;26(3):287-92. doi: 10.1097/00007632-200102010-00014. PMID 11224865
- [Background] Peng B, Zhang Y, Hou S, Wu W, Fu X. Intradiscal methylene blue injection for the treatment of chronic discogenic low back pain. Eur Spine J. 2007 Jan;16(1):33-8. doi: 10.1007/s00586-006-0076-1. Epub 2006 Feb 22. PMID 16496191
- [Background] Peng B, Pang X, Wu Y, Zhao C, Song X. A randomized placebo-controlled trial of intradiscal methylene blue injection for the treatment of chronic discogenic low back pain. Pain. 2010 Apr;149(1):124-129. doi: 10.1016/j.pain.2010.01.021. Epub 2010 Feb 18. PMID 20167430
- [Background] Levi DS, Horn S, Walko E. Intradiskal methylene blue treatment for diskogenic low back pain. PM R. 2014 Nov;6(11):1030-7. doi: 10.1016/j.pmrj.2014.04.008. Epub 2014 Apr 26. PMID 24780850
- [Background] Nguyen RT, Borg-Stein J, McInnis K. Applications of platelet-rich plasma in musculoskeletal and sports medicine: an evidence-based approach. PM R. 2011 Mar;3(3):226-50. doi: 10.1016/j.pmrj.2010.11.007. PMID 21402369
- [Background] Levi D, Horn S, Tyszko S, Levin J, Hecht-Leavitt C, Walko E. Intradiscal Platelet-Rich Plasma Injection for Chronic Discogenic Low Back Pain: Preliminary Results from a Prospective Trial. Pain Med. 2016 Jun;17(6):1010-22. doi: 10.1093/pm/pnv053. Epub 2015 Dec 26. PMID 26814283
- [Background] Tuakli-Wosornu YA, Terry A, Boachie-Adjei K, Harrison JR, Gribbin CK, LaSalle EE, Nguyen JT, Solomon JL, Lutz GE. Lumbar Intradiskal Platelet-Rich Plasma (PRP) Injections: A Prospective, Double-Blind, Randomized Controlled Study. PM R. 2016 Jan;8(1):1-10; quiz 10. doi: 10.1016/j.pmrj.2015.08.010. Epub 2015 Aug 24. PMID 26314234
- [Background] Connolly JF, Guse R, Tiedeman J, Dehne R. Autologous marrow injection as a substitute for operative grafting of tibial nonunions. Clin Orthop Relat Res. 1991 May;(266):259-70. PMID 2019059
- [Background] Muschler GF, Nitto H, Matsukura Y, Boehm C, Valdevit A, Kambic H, Davros W, Powell K, Easley K. Spine fusion using cell matrix composites enriched in bone marrow-derived cells. Clin Orthop Relat Res. 2003 Feb;(407):102-18. doi: 10.1097/00003086-200302000-00018. PMID 12567137
- [Background] Holton J, Imam M, Ward J, Snow M. The Basic Science of Bone Marrow Aspirate Concentrate in Chondral Injuries. Orthop Rev (Pavia). 2016 Sep 30;8(3):6659. doi: 10.4081/or.2016.6659. eCollection 2016 Sep 19. PMID 27761221
- [Background] Chahla J, Dean CS, Moatshe G, Pascual-Garrido C, Serra Cruz R, LaPrade RF. Concentrated Bone Marrow Aspirate for the Treatment of Chondral Injuries and Osteoarthritis of the Knee: A Systematic Review of Outcomes. Orthop J Sports Med. 2016 Jan 13;4(1):2325967115625481. doi: 10.1177/2325967115625481. eCollection 2016 Jan. PMID 26798765
- [Background] Shapiro SA, Kazmerchak SE, Heckman MG, Zubair AC, O'Connor MI. A Prospective, Single-Blind, Placebo-Controlled Trial of Bone Marrow Aspirate Concentrate for Knee Osteoarthritis. Am J Sports Med. 2017 Jan;45(1):82-90. doi: 10.1177/0363546516662455. Epub 2016 Sep 30. PMID 27566242
- [Background] Centeno CJ, Al-Sayegh H, Freeman MD, Smith J, Murrell WD, Bubnov R. A multi-center analysis of adverse events among two thousand, three hundred and seventy two adult patients undergoing adult autologous stem cell therapy for orthopaedic conditions. Int Orthop. 2016 Aug;40(8):1755-1765. doi: 10.1007/s00264-016-3162-y. Epub 2016 Mar 30. PMID 27026621
- [Background] Centeno C, Pitts J, Al-Sayegh H, Freeman M. Efficacy of autologous bone marrow concentrate for knee osteoarthritis with and without adipose graft. Biomed Res Int. 2014;2014:370621. doi: 10.1155/2014/370621. Epub 2014 Sep 7. PMID 25276781
- [Background] Pettine K, Suzuki R, Sand T, Murphy M. Treatment of discogenic back pain with autologous bone marrow concentrate injection with minimum two year follow-up. Int Orthop. 2016 Jan;40(1):135-40. doi: 10.1007/s00264-015-2886-4. Epub 2015 Jul 10. PMID 26156727
- [Background] Pettine KA, Murphy MB, Suzuki RK, Sand TT. Percutaneous injection of autologous bone marrow concentrate cells significantly reduces lumbar discogenic pain through 12 months. Stem Cells. 2015 Jan;33(1):146-56. doi: 10.1002/stem.1845. PMID 25187512
- [Background] Centeno CJ, Al-Sayegh H, Bashir J, Goodyear S, Freeman MD. A prospective multi-site registry study of a specific protocol of autologous bone marrow concentrate for the treatment of shoulder rotator cuff tears and osteoarthritis. J Pain Res. 2015 Jun 5;8:269-76. doi: 10.2147/JPR.S80872. eCollection 2015. PMID 26089699
- [Background] DePalma MJ, Ketchum JM, Saullo T. What is the source of chronic low back pain and does age play a role? Pain Med. 2011 Feb;12(2):224-33. doi: 10.1111/j.1526-4637.2010.01045.x. Epub 2011 Jan 25. PMID 21266006
- [Background] Weishaupt D, Zanetti M, Hodler J, Min K, Fuchs B, Pfirrmann CW, Boos N. Painful Lumbar Disk Derangement: Relevance of Endplate Abnormalities at MR Imaging. Radiology. 2001 Feb;218(2):420-7. doi: 10.1148/radiology.218.2.r01fe15420. PMID 11161156
- [Background] O'Neill C, Kurgansky M, Kaiser J, Lau W. Accuracy of MRI for diagnosis of discogenic pain. Pain Physician. 2008 May-Jun;11(3):311-26. PMID 18523502
- [Background] Kang CH, Kim YH, Lee SH, Derby R, Kim JH, Chung KB, Sung DJ. Can magnetic resonance imaging accurately predict concordant pain provocation during provocative disc injection? Skeletal Radiol. 2009 Sep;38(9):877-85. doi: 10.1007/s00256-009-0709-7. Epub 2009 May 9. PMID 19430778
- [Background] Carragee EJ, Don AS, Hurwitz EL, Cuellar JM, Carrino JA, Herzog R. 2009 ISSLS Prize Winner: Does discography cause accelerated progression of degeneration changes in the lumbar disc: a ten-year matched cohort study. Spine (Phila Pa 1976). 2009 Oct 1;34(21):2338-45. doi: 10.1097/BRS.0b013e3181ab5432. PMID 19755936
- [Background] Depalma MJ, Ketchum JM, Trussell BS, Saullo TR, Slipman CW. Does the location of low back pain predict its source? PM R. 2011 Jan;3(1):33-9. doi: 10.1016/j.pmrj.2010.09.006. PMID 21257131
- [Background] Levi D, Carnahan D, Horn S, Levin J. Is a History of Severe Episodic Low Back Pain an Indicator of a Discogenic Etiology? Pain Med. 2018 Jul 1;19(7):1334-1339. doi: 10.1093/pm/pnx147. PMID 29016955
- [Background] Dreyfuss P, Michaelsen M, Pauza K, McLarty J, Bogduk N. The value of medical history and physical examination in diagnosing sacroiliac joint pain. Spine (Phila Pa 1976). 1996 Nov 15;21(22):2594-602. doi: 10.1097/00007632-199611150-00009. PMID 8961447
- [Background] Ghahreman A, Ferch R, Bogduk N. The efficacy of transforaminal injection of steroids for the treatment of lumbar radicular pain. Pain Med. 2010 Aug;11(8):1149-68. doi: 10.1111/j.1526-4637.2010.00908.x. PMID 20704666
- [Background] Fairbank JC, Couper J, Davies JB, O'Brien JP. The Oswestry low back pain disability questionnaire. Physiotherapy. 1980 Aug;66(8):271-3. No abstract available. PMID 6450426
- [Background] Kolahi J, Bang H, Park J. Towards a proposal for assessment of blinding success in clinical trials: up-to-date review. Community Dent Oral Epidemiol. 2009 Dec;37(6):477-84. doi: 10.1111/j.1600-0528.2009.00494.x. Epub 2009 Sep 15. PMID 19758415
- [Background] Levi D, Horn S, Corcoran S. The Incidence of Intradiscal, Intrathecal, and Intravascular Flow During the Performance of Retrodiscal (Infraneural) Approach for Lumbar Transforaminal Epidural Steroid Injections. Pain Med. 2016 Aug;17(8):1416-22. doi: 10.1093/pm/pnv067. Epub 2015 Dec 24. PMID 26814293
- [Background] Golish SR, Hanna LS, Bowser RP, Montesano PX, Carragee EJ, Scuderi GJ. Outcome of lumbar epidural steroid injection is predicted by assay of a complex of fibronectin and aggrecan from epidural lavage. Spine (Phila Pa 1976). 2011 Aug 15;36(18):1464-9. doi: 10.1097/BRS.0b013e3181f40e88. PMID 21224775
- [Background] Kamper SJ, Ostelo RW, Knol DL, Maher CG, de Vet HC, Hancock MJ. Global Perceived Effect scales provided reliable assessments of health transition in people with musculoskeletal disorders, but ratings are strongly influenced by current status. J Clin Epidemiol. 2010 Jul;63(7):760-766.e1. doi: 10.1016/j.jclinepi.2009.09.009. Epub 2010 Jan 8. PMID 20056385
- [Background] Sharma SK, Jones JO, Zeballos PP, Irwin SA, Martin TW. The prevention of discitis during discography. Spine J. 2009 Nov;9(11):936-43. doi: 10.1016/j.spinee.2009.06.001. Epub 2009 Jul 29. PMID 19643677
- [Background] Kennedy DJ, Levin J, Rosenquist R, Singh V, Smith C, Stojanovic MP, Vorobeychik Y. Epidural Steroid Injections are Safe and Effective: Multisociety Letter in Support of the Safety and Effectiveness of Epidural Steroid Injections. Pain Med. 2015 May;16(5):833-8. doi: 10.1111/pme.12667. Epub 2015 Jan 13. PMID 25586082
- [Background] Gruber HE, Rhyne AL 3rd, Hansen KJ, Phillips RC, Hoelscher GL, Ingram JA, Norton HJ, Hanley EN Jr. Deleterious effects of discography radiocontrast solution on human annulus cell in vitro: changes in cell viability, proliferation, and apoptosis in exposed cells. Spine J. 2012 Apr;12(4):329-35. doi: 10.1016/j.spinee.2012.02.003. Epub 2012 Mar 16. PMID 22424848
- [Background] Naqvi SM, Buckley CT. Bone Marrow Stem Cells in Response to Intervertebral Disc-Like Matrix Acidity and Oxygen Concentration: Implications for Cell-based Regenerative Therapy. Spine (Phila Pa 1976). 2016 May;41(9):743-50. doi: 10.1097/BRS.0000000000001314. PMID 26630431

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT03340818/Prot_SAP_000.pdf
  • Informed Consent Form (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/18/NCT03340818/ICF_001.pdf